CLINICAL TRIAL: NCT02712658
Title: Role of K+ and Ca2+ in Development of Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Nielsen, Post.Doc, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MIK
Record Dates: First submitted 2015-10-11; First posted 2016-03-18 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Skeletal Muscle Fatigue in Humans
MeSH Terms: interventions — Terbutaline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- terbutaline (Active Comparator): terbutaline is administered by injection (0.25-0.5 mg Bricanyl, AstraZeneca diluted in 9 ml isotonic saline)
  Interventions: Drug: Terbutaline
- Placebo (Placebo Comparator): placebo is administered as isotonic saline (10 ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terbutaline — K+ transport and Ca2+ release and uptake function are stimulated by administration of terbutaline
  Arms: terbutaline
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the role of K+ and Ca2+ in development of muscle fatigue in trained young men.

ELIGIBILITY:
Inclusion Criteria:

* physical active healthy men
* aged 18-40 years

Exclusion Criteria:

* smokers
* allergy towards terbutaline
* chronic disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in time to fatigue during knee-extensor exercise | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Denmark